CLINICAL TRIAL: NCT06693427
Title: Effect of Femoral and Sciatic Nerve Blocks, Combined with General Anesthesia, in Postoperative Pain Levels and Phantom Limb Pain Development in Patients Undergoing Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: DIMITRIOS KATSAROS (Other)
Responsible Party: Sponsor-Investigator, DIMITRIOS KATSAROS, Dimitrios Katsaros, MD, G.Gennimatas General Hospital
Organization: G.Gennimatas General Hospital (Other)
Other Study IDs: GGennimatasGH 8473
Record Dates: First submitted 2024-07-24; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Phantom Limb Pain; Amputation; Anesthesia, Local
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- General Anesthesia: Patients receiving general anesthesia only.
- General Anesthesia + Blocks: Patients receiving general anesthesia and peripheral nerve blocks
  Interventions: Procedure: Peripheral Nerve Block

INTERVENTIONS:
Procedure: Peripheral Nerve Block — Femoral and Sciatic Nerve Blocks
  Groups: General Anesthesia + Blocks

SUMMARY:
The goal of this observational study is to determine the effect of femoral and sciatic nerve blocks, combined with general anesthesia, in postoperative pain levels and phantom limb pain development in patients undergoing lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower limb amputation 10cm cephalad or 10cm caudal of the knee, due to Peripheral Arterial Disease

Exclusion Criteria:

* Any form of dementia
* Prior chronic neuropathic pain as assessed with DN4 questionnaire
* Surgery under neuraxial anaesthesia
* Inability to complete a Numeric Rating Scale to assess pain
* Contraindication to ropivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for lower limb amputation 10cm cephalad or 10cm caudal of the knee, due to Peripheral Arterial Disease. All patients presented to the Emergency Department and had completed their surgery in the first 24 hours since presentation. Post-operative follow-up was every 8 hours for the first day, every 12 hours for Day 2-3. Long term follow-up was at 30 days, 3 months, 6 months and 9 months.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Presence of phantom limb pain | Total screening time up to 9 months from day of surgery (DAY 0). Timeframe: DAY 3, DAY 7, DAY 30, DAY 60, DAY 90, DAY 120, DAY 150, DAY 180, DAY 210, DAY 240, DAY 270.
  Presence of phantom limp pain and residual limp pain assessed using the Numerical Rating Scale for pain sensation (0-10, 0 being no pain, 10 being the worst imaginable pain)
Presence of phantom limb pain | Total screening time up to 9 months from day of surgery (DAY 0). Timeframe: DAY 3, DAY 7, DAY 30, DAY 60, DAY 90, DAY 120, DAY 150, DAY 180, DAY 210, DAY 240, DAY 270.
  Presence of phantom limp pain and residual limp pain assessed using the Douleur Neuropathique en 4 Questions questionnaire (total scoring 0-10, score of 4 and above indicating presence of neuropathic pain) for neuropathic pain
Presence of phantom limb pain | Total screening time up to 9 months from day of surgery (DAY 0). Timeframe: DAY 3, DAY 7, DAY 30, DAY 60, DAY 90, DAY 120, DAY 150, DAY 180, DAY 210, DAY 240, DAY 270.
  Presence of phantom limp pain and residual limp pain assessed using the painDETECT questionnaire (total scoring 0-38, 0-12 indicating an unlikely component of neuropathic pain, 13-18 an ambiguous result and 19-38 a likely component of neuropathic pain) for neuropathic pain

SECONDARY OUTCOMES:
Postoperative morphine consumption | Up to 3 days after surgery (DAY 0), i. e. until DAY 3
  All patients will be connected to an electronic pump for administration of morphine as an analgesic agent through a Patient Controlled Analgesia protocol, which enables the administration of morphine only when required by the patient. At the end of the time frame period the total morphine consumption was measured.
Postoperative pain | Up to 3 days after day of surgery (DAY 0). Assessed at: DAY 0 12 hours after end of surgery, DAY 1 , DAY 2, DAY 3
  Postoperative pain assessed using the Numerical Rating Scale for pain sensation (0-10, 0 being no pain, 10 being the worst imaginable pain)
Postoperative pain | Up to 3 days after day of surgery (DAY 0). Assessed at: DAY 0 12 hours after end of surgery, DAY 1 , DAY 2, DAY 3
  Postoperative pain assessed using the Douleur Neuropathique en 4 Questions questionnaire (total scoring 0-10, score of 4 and above indicating presence of neuropathic pain) for neuropathic pain
Postoperative pain | Up to 3 days after day of surgery (DAY 0). Assessed at: DAY 0 12 hours after end of surgery, DAY 1 , DAY 2, DAY 3
  Postoperative pain assessed using the painDETECT questionnaire (total scoring 0-38, 0-12 indicating an unlikely component of neuropathic pain, 13-18 an ambiguous result and 19-38 a likely component of neuropathic pain) for neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Katsaros, Principal Investigator — G.Gennimatas General Hospital
Locations (1):
- G. Gennimatas General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flor H. Phantom-limb pain: characteristics, causes, and treatment. Lancet Neurol. 2002 Jul;1(3):182-9. doi: 10.1016/s1474-4422(02)00074-1. PMID 12849487
- [Background] Laloo R, Ambler GK, Locker D, Twine CP, Bosanquet DC. Systematic Review and Meta-Analysis of the Effect of Perineural Catheters in Major Lower Limb Amputations. Eur J Vasc Endovasc Surg. 2021 Aug;62(2):295-303. doi: 10.1016/j.ejvs.2021.03.008. Epub 2021 Jun 2. PMID 34088614
- [Background] Geertzen J, van der Linde H, Rosenbrand K, Conradi M, Deckers J, Koning J, Rietman HS, van der Schaaf D, van der Ploeg R, Schapendonk J, Schrier E, Duijzentkunst RS, Spruit-van Eijk M, Versteegen G, Voesten H. Dutch evidence-based guidelines for amputation and prosthetics of the lower extremity: Rehabilitation process and prosthetics. Part 2. Prosthet Orthot Int. 2015 Oct;39(5):361-71. doi: 10.1177/0309364614542725. Epub 2014 Jul 24. PMID 25060393
- [Background] Karanikolas M, Aretha D, Tsolakis I, Monantera G, Kiekkas P, Papadoulas S, Swarm RA, Filos KS. Optimized perioperative analgesia reduces chronic phantom limb pain intensity, prevalence, and frequency: a prospective, randomized, clinical trial. Anesthesiology. 2011 May;114(5):1144-54. doi: 10.1097/ALN.0b013e31820fc7d2. PMID 21368651
- [Background] Alviar MJ, Hale T, Dungca M. Pharmacologic interventions for treating phantom limb pain. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006380. doi: 10.1002/14651858.CD006380.pub2. PMID 22161403
- [Background] Tilak M, Isaac SA, Fletcher J, Vasanthan LT, Subbaiah RS, Babu A, Bhide R, Tharion G. Mirror Therapy and Transcutaneous Electrical Nerve Stimulation for Management of Phantom Limb Pain in Amputees - A Single Blinded Randomized Controlled Trial. Physiother Res Int. 2016 Jun;21(2):109-15. doi: 10.1002/pri.1626. Epub 2015 Apr 1. PMID 25832306
- [Background] Horlocker TT, Vandermeuelen E, Kopp SL, Gogarten W, Leffert LR, Benzon HT. Regional Anesthesia in the Patient Receiving Antithrombotic or Thrombolytic Therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Fourth Edition). Reg Anesth Pain Med. 2018 Apr;43(3):263-309. doi: 10.1097/AAP.0000000000000763. No abstract available. PMID 29561531
- [Background] Natarajan B, Patel P, Mukherjee A. Acute Lower Limb Ischemia-Etiology, Pathology, and Management. Int J Angiol. 2020 Sep;29(3):168-174. doi: 10.1055/s-0040-1713769. Epub 2020 Jun 27. PMID 33100802
- [Background] Grant AJ, Wood C. The effect of intra-neural local anaesthetic infusion on pain following major lower limb amputation. Scott Med J. 2008 Feb;53(1):4-6. doi: 10.1258/RSMSMJ.53.1.4. PMID 18422201
- [Background] Ayling OG, Montbriand J, Jiang J, Ladak S, Love L, Eisenberg N, Katz J, Clarke H, Roche-Nagle G. Continuous regional anaesthesia provides effective pain management and reduces opioid requirement following major lower limb amputation. Eur J Vasc Endovasc Surg. 2014 Nov;48(5):559-64. doi: 10.1016/j.ejvs.2014.07.002. Epub 2014 Aug 16. PMID 25139251
- [Background] von Plato H, Peltoniemi M, Kauhanen P, Loyttyniemi E, Hamunen K, Kontinen V; FinAPain-1 study group. Combination of perineural and wound infusion after above knee amputation: A randomized, controlled multicenter study. Acta Anaesthesiol Scand. 2019 Nov;63(10):1406-1412. doi: 10.1111/aas.13440. Epub 2019 Jul 19. PMID 31281981
- [Background] Milosevic S, Strange H, Morgan M, Ambler GK, Bosanquet DC, Waldron CA, Thomas-Jones E, Harris D, Twine CP, Brookes-Howell L. Exploring patients' experiences of analgesia after major lower limb amputation: a qualitative study. BMJ Open. 2021 Dec 1;11(12):e054618. doi: 10.1136/bmjopen-2021-054618. PMID 34853109
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Lambert Aw, Dashfield Ak, Cosgrove C, Wilkins Dc, Walker Aj, Ashley S. Randomized prospective study comparing preoperative epidural and intraoperative perineural analgesia for the prevention of postoperative stump and phantom limb pain following major amputation. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):316-21. doi: 10.1053/rapm.2001.23934. PMID 11464349
- [Background] Subedi B, Grossberg GT. Phantom limb pain: mechanisms and treatment approaches. Pain Res Treat. 2011;2011:864605. doi: 10.1155/2011/864605. Epub 2011 Aug 14. PMID 22110933
- [Background] Roullet S, Nouette-Gaulain K, Biais M, Bernard N, Benard A, Revel P, Capdevila X, Sztark F. Preoperative opioid consumption increases morphine requirement after leg amputation. Can J Anaesth. 2009 Dec;56(12):908-13. doi: 10.1007/s12630-009-9185-8. Epub 2009 Nov 12. PMID 19908106
- [Background] Colvin LA, Bull F, Hales TG. Perioperative opioid analgesia-when is enough too much? A review of opioid-induced tolerance and hyperalgesia. Lancet. 2019 Apr 13;393(10180):1558-1568. doi: 10.1016/S0140-6736(19)30430-1. PMID 30983591